CLINICAL TRIAL: NCT00723515
Title: Therapeutic Effect of Two Fluoride Varnishes on White Spot Lesions: a Clinical Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pernambuco (Other)
Responsible Party: Jainara Maria Soares Ferreira, University of Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UPE 260/08
Record Dates: First submitted 2008-07-24; First posted 2008-07-28 (Estimated); Last update posted 2008-07-28 (Estimated); Status verified 2008-07

CONDITIONS: Dental Caries
Keywords: White spot lesion; Tooth remineralization; Fluoride varnishes
MeSH Terms: conditions — Dental Caries | interventions — Sodium Fluoride; sodium fluoride topical preparation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- G1 (Active Comparator): NaF (sodium fluoride varnish) with 2.26% of fluoride
  Interventions: Drug: sodium fluoride
- G2 (Experimental): NaF (sodium fluoride)2.71% of fluoride plus CaF2 (calcium fluoride)
  Interventions: Drug: sodium fluoride calcium fluoride

INTERVENTIONS:
Drug: sodium fluoride — sodium fluoride 5%
  Other Names: Duraphat®, Colgate Palmolive GmbH, Hamburg, Germany
  Arms: G1
Drug: sodium fluoride calcium fluoride — sodium fluoride 5% + calcium fluoride
  Other Names: Duofluorid XII®, FGM, Joinville, Brazil
  Arms: G2

SUMMARY:
The study hypothesis is the difference in therapeutic effect of two varnish formulations (G1 = NaF, 2.26%F, G2 = NaF, 2.71% F + CaF2). These products are commercially available in the Brazilian and international market and they are used for dental caries as white spot lesions control.

DETAILED DESCRIPTION:
The aim of this study was to evaluate the therapeutic effect of two varnish formulations (G1 = NaF, 2.26%F, G2 = NaF, 2.71% F + CaF2) on the remineralization of white spot lesions (WSL). The sample was composed of 15 (7- to 12-year-old) children with 45 active WSL in anterior permanent teeth. The children were randomly divided in two groups providing 22 lesions for G1 and 23 for G2. The children were submitted to weekly varnish applications 4 times. The WSL were evaluated twice: baseline and on week 4. Maximum lesion dimensions (mesial-distal and incisal-gingival) were measured in millimeters and classified in four grades of size. WSL were also recorded assessing lesion activity by one calibrated examiner. The Pearson chi-square and Fisher's exact tests were used (P < 0.01). WSL reductions were observed in both varnish groups (Chi-square= 0.15, d.f.=1, P=0.90); and with similar magnitude (in mm): 1.19 and 1.29 for G1 and G2, respectively. Thirty-six WLS (15 in G1 and 26 in G2) were classified as inactive in week 4 reaching an overall value of 80%. No difference was observed between G1 and G2 regarding activity scores (Fisher's exact test, p > 0.01). It can be concluded that after 4 applications the two varnish formulations tested produced similar clinical effects indicating the reduction and the control of carious activity in most WSL.

ELIGIBILITY:
Inclusion Criteria:

* regular hygiene habits (brushing teeth everyday)
* registered in public schools

Exclusion Criteria:

* dental caries such as small cavities or restorations in the target teeth (permanent anterior teeth)
* development enamel alterations (hypoplasia, fluorosis) or periodontal disease
* children using orthodontic devices
* under medical treatment
* taking any kind of medicine
* no informed consent form signed

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2007-02; Primary Completion 2007-06 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
reduction of the size of the caries lesion | 4 weeks

SECONDARY OUTCOMES:
Inactivation of carious lesions | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jainara MS Ferreira, Master, Principal Investigator — University of Pernambuco; Ana Karla R Aragão, Graduate, Study Chair — Univeristy of Pernambuco; Adriana DB Rosa, student, Study Chair — Federal University of Paraiba; Fabio C Sampaio, PhD, Study Chair — Federal Univerisity of Paraiba; Valdenice A Menezes, PhD, Study Chair — Univeristy of Pernambuco
Locations (1):
- University of Pernambuco, Camaragibe, Pernambuco, Brazil

REFERENCES:
- [Derived] Ferreira JM, Aragao AK, Rosa AD, Sampaio FC, Menezes VA. Therapeutic effect of two fluoride varnishes on white spot lesions: a randomized clinical trial. Braz Oral Res. 2009 Oct-Dec;23(4):446-51. doi: 10.1590/s1806-83242009000400015. PMID 20027453